CLINICAL TRIAL: NCT01330576
Title: Therapeutic Controlled Hypothermia in the Treatment of Neonates With Severe Necrotizing Enterocolitis
Acronym: CoolNEC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of funding
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06SG14
Record Dates: First submitted 2011-04-04; First posted 2011-04-07 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Necrotizing Enterocolitis
Keywords: Hypothermia; cooling; necrotizing enterocolitis; NEC; neonates; preterm
MeSH Terms: conditions — Enterocolitis, Necrotizing; Hypothermia; Premature Birth | interventions — Beds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard treatment of care at normothermia (Placebo Comparator): Control group: Standard treatment of care at normothermia
  Interventions: Procedure: Standard treatment of care at normothermia
- cooling blanket/mattress (Experimental): Therapeutic controlled hypothermia (33.5C) using cooling blanket/mattress
  Interventions: Procedure: cooling blanket/mattress

INTERVENTIONS:
Procedure: cooling blanket/mattress — Therapeutic controlled hypothermia (33.5C) using cooling blanket/mattress
  Arms: cooling blanket/mattress
Procedure: Standard treatment of care at normothermia — Standard treatment of care in 33.5C for 48 hours
  Arms: Standard treatment of care at normothermia

SUMMARY:
Hypothesis: Controlled hypothermia to 33.5C for 48 hours reduces the severity of critical illness in neonates with severe necrotizing enterocolitis.

ELIGIBILITY:
Inclusion Criteria:

* weight at diagnosis > 700 grams
* confirmed NEC (Bell's stage II or III)
* radiological evidence of pneumatosis coli
* systemic compromise as defined by increase in ventilation requirement and/or requiring inotopic support

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-08-02 (Actual); Primary Completion 2013-03-25 (Actual); Study Completion 2013-03-25 (Actual)

PRIMARY OUTCOMES:
Difference in sequential organ failure assessment (SOFA) score | 5 days
  Difference in sequential organ failure assessment (SOFA) score at 5 days after intervention

SECONDARY OUTCOMES:
Baseline time taken to establish full enteral feeds | 5 days
  Time to establish full enteral feeds and organ functional investigation and biomarkers at baseline, 24 hours post, 63 hours post and day 5 post intervention
Neurodevelopmental Assessment | 24 months
  Neurodevelopmental outcome with MRI at term corrected age and neurodevelopmental assessment at 3, 6,12 and 24 months and mortality data

CONTACTS AND LOCATIONS:
Locations (1):
- Great Ormond Street Hospital for Children NHS Trust, London, United Kingdom

REFERENCES:
- [Background] Hall NJ, Eaton S, Peters MJ, Hiorns MP, Alexander N, Azzopardi DV, Pierro A. Mild controlled hypothermia in preterm neonates with advanced necrotizing enterocolitis. Pediatrics. 2010 Feb;125(2):e300-8. doi: 10.1542/peds.2008-3211. Epub 2010 Jan 25. PMID 20100756